CLINICAL TRIAL: NCT00555646
Title: A Phase 2 Study of Topical PH-10 Aqueous Hydrogel and Photodynamic Therapy for the Treatment of Plaque Psoriasis
Brief Title: Topical PH-10 Aqueous Hydrogel and Photodynamic Therapy for Psoriasis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Change of dose regimen (new protocol)
Sponsor: Provectus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-10-PS-21
Record Dates: First submitted 2007-11-07; First posted 2007-11-09 (Estimated); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Each subject's study plaque areas will be assigned by the investigator to two PH-10 treatment plaque areas and one control plaque area.
  Interventions: Drug: PH-10 (rose bengal disodium 0.001%); Drug: Control

INTERVENTIONS:
Drug: PH-10 (rose bengal disodium 0.001%) — Treatment plaque area 1: PH-10 with 544 nm LED light illumination.
Drug: PH-10 (rose bengal disodium 0.001%) — Treatment plaque area 2: PH-10 with ambient light illumination.
Drug: Control — No treatment control.

SUMMARY:
This is an open label, single center, controlled study with each subject's two treatment plaque areas assigned by the investigator 1:1 to (a) PH-10 with ambient light exposure and (b) PH-10 with 544 nm LED light illumination at 10 J/cm2. A third plaque area will receive no treatment and serve as a control.

Subjects with at least three distinct, stable study plaque areas will receive the experimental therapy to two treatment plaque areas twice a week (2-5 days apart) for the lesser of 12 weeks or until remission is observed in the treatment plaque areas. If remission is observed in a treatment plaque area then treatment of that area will be discontinued and the area assessed weekly. A third plaque area (control plaque area) will receive no drug or light treatment and serve as an internal control.

Primary efficacy will be assessed 12 weeks after initial PH-10 treatment. Subjects will be followed for a total of 16 weeks to allow assessment of Durability of Response of treated lesions and comprehensive follow-up of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Stable, moderate to severe plaque psoriasis in at least three distinct plaque areas, each separated by at least a 2.5-cm band of normal skin. Study plaque areas, each covering a contiguous area up to 15 x 35 cm in size, should have a minimum plaque size of 2 cm2. All study plaque areas must be on the trunk or extremities (excluding palms, soles, scalp, and facial or intertriginous sites).
* Fitzpatrick skin type I-VI.
* Ability to understand and sign the informed consent document.

Exclusion Criteria:

* Female subjects of childbearing potential who are pregnant, attempting to conceive, or nursing an infant.
* Subjects who have received PUVA or UVB light therapy or systemic antipsoriatic therapy within 4 weeks of study treatment (two weeks for methotrexate).
* Subjects who have received topical antipsoriatic therapy (including corticosteroids, tar, anthralin, or Vitamin D analogs) to the study plaque areas within 2 weeks of study treatment.
* Subjects who have received any photosensitizing or phototoxic drug within 4 weeks of study treatment.
* Subjects who have received any approved biologic drug therapy for psoriasis within 3 months or 5 half-lives of study treatment.
* Subjects who have participated in a clinical research study within 4 weeks of study treatment.
* Subjects with a history of porphyria, systemic lupus erythematosus or xeroderma pigmentosum.
* Subjects with clinical conditions that, in the opinion of the Principal Investigator, may pose a health risk to the subject by being involved in the study or detrimentally affect regular follow-up of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Treatment Success, defined as 0 or 1 on all Psoriasis Severity Index components (erythema, induration, and scaling) and 0 or 1 on the Plaque Response scale. | 12 weeks
  Treatment Success was assessed after 12 weeks and defined as 0 or 1 on all Psoriasis Severity Index components (erythema, induration, and scaling) and 0 or 1 on the Plaque Response scale.

SECONDARY OUTCOMES:
Change in Pruritus of subject's treatment and control plaque areas using a self-assessment scale of 0-4. | 12 weeks
  Pruritus was assessed on a scale ranging from 0 (no pruritus) to 4 (frequent, troublesome pruritus that interferes with sleep or other activities).
Time to Remission (TTR) based on the (a) number of treatments and (b) days elapsed until Treatment Success is noted in each treatment plaque area. | 12 weeks
Durability of Response based on plaque areas exhibiting Treatment Success that retain this level of response. | 16 weeks
Adverse Experience. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Amir Larian, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States